CLINICAL TRIAL: NCT01717118
Title: Evaluation of Immunogenicity Levels in Women With HPV Vaccine in Mexico
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Secretaria de Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Eduardo Cesar Lazcano Ponce, Executive Director of the Center of Research in population health, Instituto Nacional de Salud Publica, Mexico
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 883
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Evaluation; Immunogenicity; Levels; Women; HPV; Vaccine; Mexico
MeSH Terms: interventions — Vaccines, Combined; human papillomavirus vaccine, L1 type 16, 18; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tetravalent Vaccine (Active Comparator): * Month 2 visit: May be scheduled on the appropriate month +/- 3 weeks.
  * Month 6, 21, 60 and 61 visit (vaccination scheme 0, 2, 6): May be programmed on the appropriate month +/- 4 weeks.
  * Month 7 and 61 visit (vaccination scheme 0, 6, 60): The time interval between the month 6/60 visit and the month 7/61 visit must be at least 3 weeks and maximum 7 weeks from the previous vaccination
  Interventions: Biological: Tetravalent Vaccine
- Bivalent Vaccine (Active Comparator): * Month 1 visit: May be scheduled 21 to 62 days after the Day 0 visit.
  * Month 6 visit: May be scheduled 161 to 216 days after the Day 0 visit.
  * Month 6 visit: The time interval between the month 6 visit and the month 7 visit must be at least 3 weeks and maximum 7 weeks from the previous vaccination.
  * Month 21, 60 and 61 visit (vaccination scheme 0, 1, 6): May be scheduled on the appropriate month +/- 4 weeks.
  * Month 61 (vaccination scheme 0, 6, 60) The time interval between the month 60 visit and the month 61 visit must be at least 3 weeks and maximum 7 weeks from the previous vaccination
  Interventions: Biological: Bivalent Vaccines

INTERVENTIONS:
Biological: Bivalent Vaccines
  Other Names: CERVARIX
  Arms: Bivalent Vaccine
Biological: Tetravalent Vaccine
  Other Names: Gardasil
  Arms: Tetravalent Vaccine

SUMMARY:
In September 2009 the National Vaccination Council approved the policy for anti-HPV vaccination in 9-year-old girls with an extended scheme of 0, 6, and 60 months, under the following justification:

* Antibody induction due to the vaccine is greater than that produced by natural exposure to the virus
* Immune response in girls 9 to 11 years of age is similar to the response obtained after three doses in women 16 to 26 years of age
* The third dose will be administered at the time when maximum protection is required, near the onset of sexual activity Thus the National Institute of Public Health was commissioned to monitor anti-HPV antibody levels in women who received the anti-HPV vaccine to determine non-inferiority of the extended scheme in 9-year-old girls compared with the traditional scheme of 3 doses in women 18 to 24 years of age. To this end, a sentinel cohort will be formed to evaluate immunogenicity levels in 3 age groups, and stratified by vaccine type. The hypothesis is that in 9-year-old girls who are administered the amplified HPV vaccination scheme (0-6-60) show immunogenicity levels that are not lower than those of adult women who have been administered the traditional scheme (0-1/2-6).

The main objectives are to monitor the levels of immunity induced by vaccination against HPV with two vaccination schemes with the quadrivalent vaccine: Traditional Extended (0-6-60 months) and traditional (0-2-6); Monitoring levels of immunity induced by vaccination against HPV with three vaccine schemes with bivalent vaccine: Extended (0-6-60 months), traditional (0-1-6) and two doses (0- 6); as well as evaluating the interchangeability of the bivalent and quadrivalent vaccines in the third dose of extended scheme. The study design is to create a sentinel cohort of women vaccinated against HPV in the following comparison groups:

* Women of nine years with extended vaccination scheme with three doses of quadrivalent vaccine (0-6-60)
* Women of nine years with extended vaccination scheme with two doses of the quadrivalent vaccine and the third dose with bivalent (0-6-60)
* Women of nine years with traditional vaccination scheme with the quadrivalent HPV vaccine (0-2-6)
* Women between 18 and 24 years with traditional vaccination scheme with the quadrivalent HPV vaccine (0-2-6)
* Women of nine years with extended vaccination scheme with three doses of bivalent vaccine (0-6-60)
* Women of nine years with extended vaccination scheme with two doses of bivalent vaccine and the third tetravalent dose
* Women of nine years with two vaccine doses scheme with the bivalent HPV vaccine (0-6)
* Women of nine years with traditional vaccination scheme with bivalent HPV vaccine (0-1-6)
* Women between 18 and 24 years with traditional vaccination scheme with bivalent HPV vaccine (0-1-6)
* To monitoring HPV infections, at month 61 of follow-up, a group of 400 women aged 14-15 years, who have not been vaccinated against HPV, will be invited , in order to make the monitoring of occurrence of HPV infections in urine per month 61, 72, 96 and 120 post dose 0 in vaccinated groups

DETAILED DESCRIPTION:
Hypothesis Girls 9 and 10 years of age who are administered the amplified anti/HPV vaccination scheme (0-6-60), show immunogenicity levels against HPV antibodies that are not lower than those of 9-year-old girls and adult women who have been administered the traditional scheme (0-1/2-6).

The vaccination schemes for HPV traditional (0-1 / 2-6) and extended (0-6-60), are equivalent from the immunologically perspective and therefore the number of memory B and T lymphocytes as well as the structure of repertoire will be not different between schemes.

Objectives The main objectives are to monitor the levels of immunity induced by vaccination against HPV with two vaccination schemes with the quadrivalent vaccine: Traditional Extended (0-6-60 months) and traditional (0-2-6); Monitoring levels of immunity induced by vaccination against HPV with three vaccine schemes with bivalent vaccine: Extended (0-6-60 months), traditional (0-1-6) and two doses (0- 6); as well as evaluating the interchangeability of the bivalent and quadrivalent vaccines in the third dose of extended scheme. The study design is to create a sentinel cohort of women vaccinated against HPV in the following comparison groups:

* Women of nine years with extended vaccination scheme with three doses of quadrivalent vaccine (0-6-60)
* Women of nine years with extended vaccination scheme with two doses of the quadrivalent vaccine and the third dose with bivalent (0-6-60)
* Women of nine years with traditional vaccination scheme with the quadrivalent HPV vaccine (0-2-6)
* Women between 18 and 24 years with traditional vaccination scheme with the quadrivalent HPV vaccine (0-2-6)
* Women of nine years with extended vaccination scheme with three doses of bivalent vaccine (0-6-60)
* Women of nine years with extended vaccination scheme with two doses of bivalent vaccine and the third tetravalent dose
* Women of nine years with two vaccine doses scheme with the bivalent HPV vaccine (0-6)
* Women of nine years with traditional vaccination scheme with bivalent HPV vaccine (0-1-6)
* Women between 18 and 24 years with traditional vaccination scheme with bivalent HPV vaccine (0-1-6)
* To monitoring HPV infections, at month 61 of follow-up, a group of 400 women aged 14-15 years, who have not been vaccinated against HPV, will be invited , in order to make the monitoring of occurrence of HPV infections in urine per month 61, 72, 96 and 120 post dose 0 in vaccinated groups

Methodology

Study design:

Creating a sentinel cohort of women vaccinated against HPV in three comparison groups:

* Women of nine years with extended vaccination scheme with three doses of quadrivalent vaccine (0-6-60)
* Women of nine years with extended vaccination scheme with two doses of the quadrivalent vaccine and the third dose with bivalent (0-6-60)
* Women of nine years with traditional vaccination scheme with the quadrivalent HPV vaccine (0-2-6)
* Women between 18 and 24 years with traditional vaccination scheme with the quadrivalent HPV vaccine (0-2-6)
* Women of nine years with extended vaccination scheme with three doses of bivalent vaccine (0-6-60)
* Women of nine years with extended vaccination scheme with two doses of bivalent vaccine and the third tetravalent dose
* Women of nine years with two vaccine doses scheme with the bivalent HPV vaccine (0-6)
* Women of nine years with traditional vaccination scheme with bivalent HPV vaccine (0-1-6)
* Women between 18 and 24 years with traditional vaccination scheme with bivalent HPV vaccine (0-1-6) Selecting the study population.

A fraction of the population of females will be invited to participate in the study proportionately, combining strategies in schools and the community.

A total of 2450 women will be recruited. For the study purposes, they will be classified by vaccine type administered, (tetravalent and bivalent), as well as by age group and vaccination scheme.

Forming groups for evaluation.

Two groups of participants will be formed. Participants will be classified by vaccine type received:

1. Bivalent Vaccine. This group will consist of a total of 2000 women. Two thirds of them will be 9 to 10 years of age, and 500 will be 18 to 24 years of age. In the first age group, 1000 of them will be administered the vaccine in the amplified scheme of 0, 6, 60 months. Five hundred females from this age group will be administered the vaccine according to the traditional scheme of 0, 1, 6 months. All females from the 18 to 24 age group will be administered the traditional scheme of 0, 1, 6 months.
2. Tetravalent Vaccine:

A total of 450 females will participate. The 9 to 10 year age group will include 300 women, and the 18 to 24 year age group will include 150 females.

The vaccination scheme will be conformed as follows: In the group of 9- to 10-year-olds, 150 of them will be administered the vaccine in the amplified scheme of 0, 6, 60 months, and the remaining 150 will receive the vaccine under the traditional scheme of 0, 2, 6 months. The group of 18- to 24-year-old women will be conducted under the traditional scheme of 0, 2 and 6 months.

The vaccination scheme will be assigned according to number in the record and/or geographical location.

For quantification of immunological memory of B and T lymphocytes and characterizing lymphocytes B repertoire in women vaccinated against HPV, 60 participants for group, recruited for medical evaluation at month 60.

To evaluate the interchangeability of quadrivalent and bivalent vaccines a randomization will be performed in the group of girls aged 14-15 years who have been assigned at the beginning of the project with extended vaccination scheme (0-6-60) with the bivalent vaccine, so that one third of this group will receive the bivalent vaccine, another third will receive the quadrivalent vaccine and the remaining third will no longer receive additional doses.

ELIGIBILITY:
Inclusion Criteria:

* • Women 18 to 24 years of age who agree to participate by signing an informed consent form prior to recruitment.

  * Girls 9 and 10 years of age whose father/mother/guardian signs the informed consent form to participate in the study.

Exclusion Criteria:

* • Prior administration of an anti-HPV vaccine

  * Pregnant women or women planning to get pregnant in the next 8 months.
  * Auto-immune diseases
  * Women with a history of Guillain Barré syndrome.
  * Prior administration of immunoglobulins and/or any blood product in the past 6 months before the study's first vaccine dose.

Ages: 9 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000 (Actual)
Dates: Start 2009-11; Primary Completion 2015-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
To monitor immunogenicity levels induced by anti/HPV vaccine in traditional squeme | 6 months
  Bivalent Vaccine: Five hundred females from this age group will be administered the vaccine according to the traditional scheme of 0, 1, 6 months. All females from the 18 to 24 age group will be administered the traditional scheme of 0, 1, 6 months.
  Tetravalent Vaccine:
  150 will receive the vaccine under the traditional scheme of 0, 2, 6 months. The group of 18- to 24-year-old women will be conducted under the traditional scheme of 0, 2 and 6 months.

SECONDARY OUTCOMES:
To monitor immunogenicity levels induced by anti/HPV vaccine in extended squeme | 60 months
  BIVALENT VACCINE: This group will consist of a total of 2000 women. Two thirds of them will be 9 to 10 years of age, and 500 will be 18 to 24 years of age. In the first age group, 1000 of them will be administered the vaccine in the amplified scheme of 0, 6, 60 months.
  TETRAVALENT VACCINE: the group of 9- to 10-year-olds, 150 of them will be administered the vaccine in the amplified scheme of 0, 6, 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo C Lazcano, Phd, MD, Principal Investigator — National Institute of Public Health Mexico; Aurelio Cruz, Valdez, Study Director — National Institute of Public Health Mexico; Janet L. Pacheco, Study Chair — National Institute of public Health
Locations (1):
- Centro Médico Cuauhtemoc, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Lazcano-Ponce E, Torres-Ibarra L, Cruz-Valdez A, Salmeron J, Barrientos-Gutierrez T, Prado-Galbarro J, Stanley M, Munoz N, Herrero R, Hernandez-Avila M. Persistence of Immunity When Using Different Human Papillomavirus Vaccination Schedules and Booster-Dose Effects 5 Years After Primary Vaccination. J Infect Dis. 2019 Jan 1;219(1):41-49. doi: 10.1093/infdis/jiy465. PMID 30085139
- [Derived] Lazcano-Ponce E, Stanley M, Munoz N, Torres L, Cruz-Valdez A, Salmeron J, Rojas R, Herrero R, Hernandez-Avila M. Overcoming barriers to HPV vaccination: non-inferiority of antibody response to human papillomavirus 16/18 vaccine in adolescents vaccinated with a two-dose vs. a three-dose schedule at 21 months. Vaccine. 2014 Feb 3;32(6):725-32. doi: 10.1016/j.vaccine.2013.11.059. Epub 2013 Dec 16. PMID 24355090